CLINICAL TRIAL: NCT06173739
Title: The Effect of Peri-Implant Soft Tissue Phenotype on the Severity of Peri-Implant Diseases and the Outcomes of Non-Surgical Mechanical Treatment
Brief Title: Peri-implant Phenotype, Calprotectin and Mmp-8 Levels in Cases Diagnosed With Peri-implant Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beliz Önder (Other)
Responsible Party: Sponsor-Investigator, Beliz Önder, Assistant Professor, Bilecik Seyh Edebali Universitesi
Organization: Bilecik Seyh Edebali Universitesi (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BSEU-ONDER-001
Record Dates: First submitted 2023-11-24; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: peri-implant disease; calprotectin; phenotype
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peri-implant mucositis (Active Comparator): It is defined as widespread inflammatory disease of the soft tissue surrounding endosseous implants without loss of crestal bone or marginal bone. Peri-implant mucositis is diagnosed by pain, swelling, redness and bleeding on probing in the soft tissue around the dental implant.
  Diagnosis will be completed based on radiographic and clinical findings at the first encounter with the patient.
  In the second session, PICF (peri-implant crevicular fluid) will be collected from both groups of implants and phenotype evaluations will be made.
  Following the recording of clinical parameters (PD, GI, PI, CAL, BOP), non-surgical mechanical treatment will be applied to both groups.
  Interventions: Procedure: Non-surgical mechanical treatment
- Peri-implantitis (Active Comparator): Peri-implantitis is a pathology that occurs in the tissues around dental implants, characterized by inflammation of the peri-implant mucosa and destruction of marginal and crestal bone. Clinical diagnosis is defined by the presence of bleeding on probing, the presence of pathological pockets, exudate, swelling, edema, and hyperemia, while findings of bone loss are supported by radiography.
  Diagnosis will be completed based on radiographic and clinical findings at the first encounter with the patient.
  In the second session, PICF (peri-implant crevicular fluid) will be collected from both groups of implants and phenotype evaluations will be made.
  Following the recording of clinical parameters (PD, GI, PI, CAL, BOP), non-surgical mechanical treatment will be applied to both groups.
  Interventions: Procedure: Non-surgical mechanical treatment

INTERVENTIONS:
Procedure: Non-surgical mechanical treatment — Nonsurgical mechanical therapy (NSMT) aims to control infection and minimize bacterial burden through debridement of the implant surface. It is the gold standard treatment method for both peri-implantitis and peri-implant mucositis.
  Non-surgical mechanical treatment will be applied to patients with the purpose of surface debridement and reducing bacterial flora in implants with peri-implant disease for which clinical examination has been completed and the diagnosis has been confirmed. All intraoral implants of the patients will be evaluated and all implants that do not meet the clinical definition of health will be intervened. Each implant surface will be treated with a titanium curette. In all groups, mechanical debridement was performed on the surfaces by the same clinician.
  The procedure will continue gently until it is felt that it has been adequately debrided. Subgingival irrigation will be performed with physiological saline. Post NSMT No medication will be administered.

SUMMARY:
Following the implantation procedures; The peri-implant mucosa may begin to show signs of inflammation depending on the patient (bruxism, lack of oral hygiene) or other factors (planning errors, iatrogenic factors). These signs of inflammation may remain limited to soft tissue or may progress to bone depending on the host response. Another relevant factor in such cases is peri-implant mucosa thickness. Our study aims to investigate the effect of peri-implant soft tissue thickness on the degree of peri-implant disease and the contribution of soft tissue augmentation procedures applied with subepithelial connective tissue graft and non-surgical mechanical treatment results, accompanied by clinical and biochemical parameters.

DETAILED DESCRIPTION:
The study was carried out in Van Yüzüncü Yıl University Faculty of Dentistry, in patients who were diagnosed with inflammation or bone loss around their implants and were referred to Periodontology Department for the treatment of the relevant areas, aged between 18-65, systemically healthy, non-smokers, and without any drug allergies. and will be conducted on 50 volunteer individuals who do not require advanced surgical techniques. The peri-implant soft tissue phenotype of all participants who are detected to have peri-implant disease and will be included in the study will be measured, necessary clinical and radiological examinations will be performed, necessary samples will be collected and conventional mechanical treatments will be applied. The data of all participants will be collected again in the 6th month following the treatment. Study details are given below: Patients who will participate in the study will be explained the details of the application and the research to be conducted and will have to sign an informed consent form.

Detailed anamnesis of patients who meet the selection criteria will be taken and clinical and radiological examinations will be performed. Patients with caries on their teeth will be directed to Restorative Dentistry Department and restorations of existing caries will be made at the relevant clinic. Patients will be given oral hygiene training before the mechanical treatment of peri-implant diseases.

Peri-implant crevice fluid (PICF) samples will be collected before mechanical treatment of the diseased implant areas of individuals is initiated. The areas will be isolated from saliva with cotton pellets, dried with light air, and the paper strips will be kept in the trough for 30 seconds. Paper strips obtained from each implant will be placed in Eppendorf tubes containing isotonic Ph:7.4 phosphate buffer solution and stored at -40 ° C until analyzed in the laboratory department of our clinic.

Routine periodontal parameters such as plaque index, gingival index, bleeding on probing, probing pocket depth, and clinical attachment level of the individuals whose PICF samples are collected will be measured and recorded with the help of Williams-type plastic probes.

Following these procedures, the patients; peri-implant phenotype will be evaluated. In the evaluation, the traditional transgingival probing technique and a newly developed technique will be used simultaneously and their correlations with each other will be examined. In the transgingival probing technique, measurements will be made from two points: apical of the free gingival groove and coronal of the mucogingival composition. After the peri-implant mucosa thickness measurement points are determined with a marker pen, Xylocaine® spray (Vemcaine 10%, lidocaine) or, if necessary, local anesthetic (Maxicaine, lidocaine hydrochloride) will be applied to prevent the patient from feeling pain. Measurements will be made from the marked points in a direction perpendicular to the peri-implant mucosa, using a 10-gauge endodontic spreader (G-Star Medical Co., Ltd., Guangdong, China) with a silicone stopper until its contact with the alveolar bone is felt. Since excessive force will cause the spreader to exceed the soft tissue and advance in the alveolar bone, care should be taken to apply only light forces that can be limited to the soft tissue. After all measurements are repeated twice by the same researcher at 10-minute intervals, the amount of peri-implant mucosa thickness in each region will be determined by taking the average of the two measurements. If the millimetric values obtained as a result of measurements are less than 1 mm, thin phenotype; If it is more than 1 mm, it will be classified as thick phenotype. The second gingival phenotype evaluation in individuals with peri-implant disease will be performed with the Hu-Friedy Colorvue Biotip Probe®, a newly developed probe with a colored tip that will be placed in the peri-implant pocket. The white probe will first be placed in the peri-implant pocket with a pressure of less than 25 N. If the color of the probe reflects from the gingival tissue, the phenotype will be recorded as thin. If the white color is not visible, the green probe will be placed in the pocket in the same way and if the color is reflected, the phenotype will be classified as medium thickness. If the Green tip is not visible through the gingival tissue, the Blue probe will be used and if the only color seen is Blue, the phenotype will be classified as thick. If blue is not visible, the peri-implant mucosa tissue will be recorded as too thick.

Then, traditional mechanical debridement with titanium curettes will be applied to areas with peri-implant disease. The area will be irrigated with physiological saline from time to time. Following the procedure, patients will be called for control at the 1st, 3rd and 6th months. Oral hygiene instructions will be repeated when necessary. At the 6th month, all clinical parameters examined will be measured again and PICF samples will be collected again.

All procedures will be performed by the same researcher. After the target number of patients is reached, the PICF samples collected will be sent to the laboratory for analysis using ELISA (Enzyme-linked immunosorbent assay) kits. Statistical analysis will be performed and interpreted for the features emphasized.

ELIGIBILITY:
Inclusion Criteria:

* -Systemically healthy,
* Non-smoker,
* There is no drug allergy and no advanced surgical techniques are required.
* 39 volunteers, aged 18-65, who applied to the Department of Periodontics with complaints of infection around the implant or were referred to our clinic, will be included.

Exclusion Criteria:

* Any drug allergy,

  * Pregnant or breastfeeding,
  * smoker
  * Having a systemic disability,
  * Peri-implant disease requiring advanced surgical techniques for treatment
  * Individuals who are not volunteers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Probing Depth(PD) | Immediately before procedure
  The depth of the peri-implant pocket or groove was measured with a plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland) from 4 regions of the peri-implant mucosa: mesial, distal, lingual/palatinal and buccal. No extra force was applied to the plastic probe during measurement. The probe placed in the pocket was held parallel to the abutment with a force equal to its own weight (approximately 0.25 N). At the point where resistance is felt at the bottom of the pocket without losing contact with the implant surface; The value corresponding to the margin was recorded on the plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland). All measurement values were collected and averaged, and the average probing depth of the relevant implant was determined.
Probing Depth(PD) | After 6 months procedure
  The depth of the peri-implant pocket or groove was measured with a plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland) from 4 regions of the peri-implant mucosa: mesial, distal, lingual/palatinal and buccal. No extra force was applied to the plastic probe during measurement. The probe placed in the pocket was held parallel to the abutment with a force equal to its own weight (approximately 0.25 N). At the point where resistance is felt at the bottom of the pocket without losing contact with the implant surface; The value corresponding to the margin was recorded on the plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland). All measurement values were collected and averaged, and the average probing depth of the relevant implant was determined.
Gingival Index (GI) | Immediately before procedure
  The plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland) is placed in the groove or pocket without pressure.
  bleeding from 4 regions (mesial, distal, lingual/palatinal and buccal) scoring was done. The gingival index score for the relevant implant is the total value Obtained by taking the average. Gingival index, inflammation in the peri-implant mucosa is one of the important indicators.
Gingival Index (GI) | After 6 months procedure
  The plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland) is placed in the groove or pocket without pressure.
  bleeding from 4 regions (mesial, distal, lingual/palatinal and buccal) scoring was done. The gingival index score for the relevant implant is the total value Obtained by taking the average. Gingival index, inflammation in the peri-implant mucosa is one of the important indicators.
Plaque Index(PI) | Immediately before procedure
  The area around the abutment to be measured was isolated with cotton pads and gently dried with air-water spray.
  Plaque was collected from around the groove or pocket with the help of a plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland).
Plaque Index(PI) | After 6 months procedure
  The area around the abutment to be measured was isolated with cotton pads and gently dried with air-water spray.
  Plaque was collected from around the groove or pocket with the help of a plastic probe (KERR- Hawe Caliber Plastic Periodontal Probe, Switzerland).
Bleeding on Probing (BOP) | Immediately before procedure
  The bleeding on probing score is the gold standard for detecting peri-implant diseases. If bleeding occurs after the probe is placed in the pocket, it is scored as positive (+), otherwise it is scored as negative (-).
Bleeding on Probing (BOP) | After 6 months procedure
  The bleeding on probing score is the gold standard for detecting peri-implant diseases. If bleeding occurs after the probe is placed in the pocket, it is scored as positive (+), otherwise it is scored as negative (-).
Clinical Attachment Level (CAL) | Immediately before procedure
  CAL; It is defined as the distance from the cemento-enamel junction (CEJ) on tooth surfaces to the apical of the pocket base. In the presence of gingival recession; The gingival margin migrates apical to the CEJ. In this case, CAL; length of gingival recession and probing It is calculated as the sum of the depth.
Clinical Attachment Level (CAL) | After 6 months procedure
  CAL; It is defined as the distance from the cemento-enamel junction (CEJ) on tooth surfaces to the apical of the pocket base. In the presence of gingival recession; The gingival margin migrates apical to the CEJ. In this case, CAL; length of gingival recession and probing It is calculated as the sum of the depth.
Calprotectin (CAL) | Immediate before procedure
  PICFs collected from the peri-implant margin with paper strips are analyzed by ELISA method. In this method, the amount of CLP, a degradation protein, is calculated. CLP is an antimicrobial protein and inflammation marker.
Calprotectin (CAL) | After 6 months procedure
  PICFs collected from the peri-implant margin with paper strips are analyzed by ELISA method. In this method, the amount of CLP, a degradation protein, is calculated. CLP is an antimicrobial protein and inflammation marker.
Matrix Metalloproteinaz-8(MMP-8) | Immediate before procedure
  PICFs collected from the peri-implant margin with paper strips are analyzed by ELISA method. MMP-8 is currently used in the prediction, diagnosis, treatment prognosis and treatment of periodontal disease.
  It is considered one of the main biomarkers used for classification. On the other hand, effective periodontal treatment and MMP inhibitor adjuvant drugs are effective in the progression of periodontal disease by reducing the MMP-8 level in GCF (gingival crevicular fluid) and saliva.
  It has been shown to have inhibitory effects. Collagenase, which also plays a role in inflammation of peri-implant connective tissue, and gelatinases, with high levels of MMP-8 in peri-implant crevice fluid. has been associated. Low MMP-8 level was determined to indicate peri-implant health, while high regulation of MMP 8 showed inflammation.
Matrix Metalloproteinaz-8(MMP-8) | After 6 months procedure
  PICFs collected from the peri-implant margin with paper strips are analyzed by ELISA method. MMP-8 is currently used in the prediction, diagnosis, treatment prognosis and treatment of periodontal disease.
  It is considered one of the main biomarkers used for classification. On the other hand, effective periodontal treatment and MMP inhibitor adjuvant drugs are effective in the progression of periodontal disease by reducing the MMP-8 level in GCF (gingival crevicular fluid) and saliva.
  It has been shown to have inhibitory effects. Collagenase, which also plays a role in inflammation of peri-implant connective tissue, and gelatinases, with high levels of MMP-8 in peri-implant crevice fluid. has been associated. Low MMP-8 level was determined to indicate peri-implant health, while high regulation of MMP 8 showed inflammation.

SECONDARY OUTCOMES:
Peri-implant phenotype | Before non-surgical mechanical treatment
  While evaluating the peri-implant tissue phenotype, peri-implant mucosa dimensions include keratinized tissue width, mucosa thickness and supracrestal tissue height; Bone level is also included in the phenotype elements.
  When measuring keratinized gums; Williams probe was used. While determining the biotype, Hu-Friedy Colorvue probes were used. Mucosa thickness is; Transgingival probing measurement technique was used. Supracrestal tissue height was measured by transmucosal probing.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Unıversity, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared during the publication phase.

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S313-S318. doi: 10.1002/JPER.17-0739. PMID 29926955

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT06173739/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT06173739/ICF_001.pdf